CLINICAL TRIAL: NCT06434259
Title: Long-term Results of an Interactive Mobile Health Support System and Daily Home-weighing as an add-on to Pediatric Obesity Lifestyle Treatment: A 3-year Pragmatic Clinical Trial
Brief Title: Evaluation of Long-term Digital Childhood Obesity Treatment
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal Investigator, Karolinska Institutet
Other Study IDs: Evira100
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Childhood Obesity; Treatment Adherence
Keywords: Mobile Health; Support System; Behavioral Treatment; Self-Monitoring
MeSH Terms: conditions — Pediatric Obesity; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digi-physical treatment group: Usual care (behavioral treatment) plus the support system for self- monitoring of weight and communication with the clinic during three years of treatment.
  Interventions: Device: Digi-physical support system
- Control group: Children treated with usual care according to regular treatment routines registered in the Swedish childhood obesity treatment register, BORIS

INTERVENTIONS:
Device: Digi-physical support system — A support system named Evira will be used to provide behavioral treatment.
  Groups: Digi-physical treatment group

SUMMARY:
This study aims to evaluate if a web-based digital support system aiming to replacing or complement standardized pediatric behavioural obesity treatment. The hypothesis is that a digital system of communication between the family and the clinic can generate improved treatment results (change in BMI SDS) and reduce the number of missed visits.

DETAILED DESCRIPTION:
Childhood obesity treatment is time consuming for both the health care system, and for the involved families. There is an association between the intensity and the outcome of treatment.

In this study all children who start treatment for childhood obesity will use a digital support system as a complement to behavioral treatment. The digital support system includes daily weighing on scales that do not show any digits, linked to a mobile app where weight development is shown as a moving average in the form of BMI standard deviation score (SDS). The app also provides an individual target curve visualizing the expected weight journey. Weight in growing children is complex to interpret why BMI SDS is used. Objective data from scale are automatically transferred to the database and the clinic and the family have direct contact with the clinic via the app.

The present study is a continuation of the investigators previous one-year study, Clinicaltrials.gov ID: NCT04323215. In this follow-up study, the investigators aim to assess the treatment outcomes over a three-year period.

The evaluation will be carried out on 107 children who underwent digi-physical treatment for three years. The results will be compared with a matched control group (n=321) from the Swedish childhood obesity treatment register, BORIS.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)

Exclusion Criteria:

* None

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children who start treatment for childhood obesity at Martina children Hospital will use a digital support system as a complement to behavioral treatment. 107 children in the digit-physical group and 321 children in the control group, aged 4-17.9 years, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in degree of obesity | From start of treatment to three years follow-up
  Measured by BMI standard deviation score. Digi-physical group vs. control group

SECONDARY OUTCOMES:
The use of the support system - weighings | From start of treatment to three years follow-up
  Number of weighings/week
The use of the support system - text messages | From start of treatment to three years follow-up
  Number text messages/week
Number of physical visits | From start of treatment to three years follow-up
  Visits to the clinic. Digi-physical group vs. control group
Number of cancelation of physical visits | From start of treatment to three years follow-up
  Visits to the clinic. Digi-physical group vs. control group
Number of patients not showing up to physical visit | From start of treatment to three years follow-up
  Visits to the clinic. Digi-physical group vs. control group

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson Liljeqvist, PhD, Principal Investigator — Karolinska Institutet, CLINTEC, Division of pediatrics
Locations (1):
- Childrens Hospital Martina, Stockholm, Sweden

REFERENCES:
- [Result] Hagman E, Johansson L, Kollin C, Marcus E, Drangel A, Marcus L, Marcus C, Danielsson P. Effect of an interactive mobile health support system and daily weight measurements for pediatric obesity treatment, a 1-year pragmatical clinical trial. Int J Obes (Lond). 2022 Aug;46(8):1527-1533. doi: 10.1038/s41366-022-01146-8. Epub 2022 May 31. PMID 35641569